CLINICAL TRIAL: NCT01752452
Title: Effect of Ulnar Styloid Fracture on the Outcome of Distal Radial Fractures Treated With External Fixation
Status: Completed | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yi-xin Chen, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: BE20116003
Record Dates: First submitted 2012-12-11; First posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Fracture of Distal End of Radius; Fracture of Ulnar Styloid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Untreated ulnar styloid fracture may affect the outcomes of distal radial fracture patient treated with external fixation.

ELIGIBILITY:
Inclusion Criteria:

* unstable distal radial fracture
* fixed with external fixator

Exclusion Criteria:

* multiple fracture
* open fracture
* nerve injury
* vascular injury

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unstable distal radial fracture patients: (1) the initial dorsal angulation >20°, (2) with dorsal or volar comminution of the metaphysis, (3) shortening of radius >5 mm, and (4) with an associated ulnar fracture.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2009-01; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
wrist motion range | 3 months, 6 months, and 1 year
  extension, flexion, radial deviation, ulnar deviation, forearm pronation and forearm supination
ulnar sided pain | 3 months, 6 months, and 1 year
  presence of ulnar-sided wrist pain during daily activities was recorded

SECONDARY OUTCOMES:
radiographic analysis | 6 weeks, 3 months, and 1 year
  Standard anterior-posterior and lateral radiographs were obtained at each time point to evaluate fracture healing and the alignment of the distal part of the radius. Radial inclination, volar tilt, and radial height were measured

CONTACTS AND LOCATIONS:
Overall Officials: Yi-xin Chen, M.D., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China